CLINICAL TRIAL: NCT05851248
Title: Free Mucogingival Graft for Isolated Root Coverage and Correct Unfavorable Mucogingival Conditions in Lower Incisors: a Randomized Clinical Trial
Brief Title: Free Mucogingival Graft for Isolated Root Coverage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Antonio José Ortiz Ruiz, MD, Professor and Researcher, Universidad de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4157/2022
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Free Mucogingival Grafts; Gingival Recession; Root Coverage; Periodontal Plastic Surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Buccal muco-gingival tissue graft (Experimental)
  Interventions: Procedure: Buccal muco-gingival tissue graft
- Palatal connective tissue graft (Active Comparator)
  Interventions: Procedure: Palatal connective tissue graft

INTERVENTIONS:
Procedure: Buccal muco-gingival tissue graft — Recipient Site Preparation. In the GR, a sulcular incision limited to the vestibular face will be made, which will continue until reaching the tip of the buccal papillae on each side of the GR. Two vertical incisions from the base of the two papillae to the bottom of the vestibule and one horizontal incision will connect the ends of both vertical incisions to remove the pedicle tissue. The exposed root surface will be cleaned and smoothed with mini-curettes.
  Donor site preparation. The incisions will be made in the same way as in the recipient area, including both papillae. The vertical incision will measure the distance from the cementoenamel junction (CEJ) to the bony dehiscence in the GR tooth, plus at least 2 mm. The tissue between the incisions will be elevated fjull or partial thickness close to the bone in the keratinized portion and superficially in the mucosal portion. A soft tissue substitute will be adapted and sutured to protect the donor site.
  Arms: Buccal muco-gingival tissue graft
Procedure: Palatal connective tissue graft — Recipient Site Preparation. In the GR, a sulcular incision limited to the vestibular face will be made, which will continue until reaching the tip of the buccal papillae on each side of the GR. Two vertical incisions from the base of the two papillae to the bottom of the vestibule and one horizontal incision will connect the ends of both vertical incisions to remove the pedicle tissue. The exposed root surface will be cleaned and smoothed with mini-curettes.
  Donor site preparation A connective tissue graft will be taken from the palatal area, at the level of the premolars, which will include the two papillae. The size of the graft will be the same as that of the recipient area. A soft tissue substitute will be adapted and sutured to protect the donor site, especially if there is exposed bone.
  Arms: Palatal connective tissue graft

SUMMARY:
The goal of this clinical trial is to to describe and evaluate an approach, free mucogingival graft (FMG), in periodontal plastic surgery for root coverage (RC) in lower incisor gingival recessions (GR) with mucogingival conditions and deformities (MCD) that might negatively influence the outcomes of conventional RC procedures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients with deep GR associated with lower incisor MCD.
* Full mouth plaque and bleeding scores were <20%.

Exclusion Criteria:

Patient characteristics:

* Smoking ≥10 cigarettes a day.
* Medications or systemic contraindications for oral surgery.
* Pregnancy.

Defects:

* Thin scalloped biotype (AND/OR)
* Underlying bone dehiscence (AND /OR)
* Generalized GR affecting most sextants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-04-22 (Estimated)

PRIMARY OUTCOMES:
buccal Recession (bREC) | 12 months
  Buccal recession measurement, will be assessed with a periodontal probe, measured in mmm on the buccal aspect, from the CEJ to the gingival margin zenith.

SECONDARY OUTCOMES:
buccal Clinical Attachment Level (bCAL) | 12 months
  bCAL will be assessed with a periodontal probe, measured in mm from the CEJ to the bottom of the pocket, on the buccal aspect.
interproximal Clinical Attachment Level (iCAL) | 12 months
  iCAL will be assessed with a periodontal probe, measured in mm from the CEJ to the bottom of the pocket, on the interproximal aspect.
Interproximal papilla tip location (PT) | 12 months
  Taking as reference the level of the mid-axis of the tooth, PT will be measured the distance from the CEJ at the zenith of the tooth to the tip of the papilla. A positive value will be recorded when the tip of the papillae is located coronally to the CEJ and a negative value otherwise.
  This outcome will be assessed with a periodontal probe and measured in mmm.
keratinized tissue width (KT) | 12 months
  KT will be assessed with a periodontal probe, measured in mm on the buccal aspect, from the gingival margin to the mucogingival line.
vestibule depth (VD) | 12 months
  VD will be measured, from the mucosal margin to the point of greatest concavity of the mucobuccal fold. The measure will be assessed with a periodontal probe in mm.
Soft tissue attached to alveolar bone (STAB) | 12 months
  STAB will be measured from the gingival margen to the perpendicular mucosal insertion. The measure will be assessed with a periodontal probe in mm.

OTHER OUTCOMES:
Root Coverage (RC percentage) | 12 months
  RC percentage will be calculated by the following formula: [(basaline recession depth - 12 months recession depth) / basaline recession depth] x100. The measure will be assessed with a periodontal probe in mm.
Complete root coverage (CRC) | 12 months
  It will assessed if the gingival margen is at or above the CEJ. The measure will be assessed with a periodontal probe in mm.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Odontologico Del Sureste Slp, Murcia, Murcia, Spain